CLINICAL TRIAL: NCT05412147
Title: A Pilot Study of the Effect of RECO-18 Containing Natural Plant Extracts on Infertile Women Undergoing in Vitro Fertilization-embryo Transfer
Brief Title: The Effect of RECO-18 on Infertile Women Undergoing in Vitro Fertilization-embryo Transfer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-KY-063
Record Dates: First submitted 2022-05-24; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-04

CONDITIONS: Fertility Disorders; Infertility, Female
Keywords: pregnancy rate; in vitro fertilization-embryo transfer
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): The control group takes the multi-vitamins (Elevit, Bayer S.A.) with the dosage of one tablet per day on the 1st to 5th day of menstruation, then perform ovulation induction on the second menstrual cycle, and continue to take multi-vitamins until the day of oocyte retrieval.
  Interventions: Dietary Supplement: Multi-vitamins
- Treatment group (Experimental): The treatment group begins to take Reco-18 on the 1st to 5th day of menstruation with a dosage of 4 pills per day for the whole menstrual cycle, then perform ovulation induction on the second menstrual cycle, and continue to take Reco-18 until the day of oocyte retrieval.
  Interventions: Dietary Supplement: RECO-18

INTERVENTIONS:
Dietary Supplement: RECO-18 — 4 pills daily, oral
  Arms: Treatment group
Dietary Supplement: Multi-vitamins — one tablet daily, oral
  Arms: Control group

SUMMARY:
How to improve the fertility of infertile women has become a hot topic in the field of assisted reproduction. Animal experiment has shown that RECO-18 significantly improved the female fertility in mice, and the specific mechanism was related to reducing follicular atresia, promoting follicle development and improving oocyte quality. Therefore the investigators aim to conduct a pilot study to explore the effect of RECO-18 in infertile women undergoing assisted reproduction treatment. This study is a prospective, randomized, controlled clinical study. The treatment group takes RECO-18 while the control group takes the multi-vitamins. The primary indicator is the ongoing pregnancy rate at 12 weeks' gestation; the secondary indicators are the number of oocytes retrieved, the normal fertilization rate and the rate of high quality embryos, implantation rate, clinical pregnancy rate, and early miscarriage rate.

DETAILED DESCRIPTION:
Mitochondrial function is closely related to oocyte quality in female. Deficiency of multiple micronutrients is common in infertile women, and supplementation with multiple micronutrients has antioxidant effects to reduce the damage of oxidative stress to fertility, and helps to improve the outcomes of assisted reproductive treatment. RECO-18 is a functional food containing a variety of plant extracts and enzymatic soy phospholipids. In in vivo and in vitro senescent models, the investigators found RECO-18 to improve oocyte quality mainly by regulating the mitochondrial apoptosis pathway. The investigators also found RECO-18 significantly improved the fertility of mice, and the specific mechanism was related to reducing follicular atresia, promoting follicle development and improving oocyte quality. Based on the animal experiments, the investigators intend to conduct a clinical trial to explore whether RECO-18 plays a role in improving oocyte and embryo quality and pregnancy outcomes in infertile women undergoing in vitro fertilization-embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* female, 20 to 40 years old
* the 1st or 2nd cycle of IVF/ICSI treatment
* BMI≤30Kg/m2
* with bilateral ovaries
* be eligible for IVF/ICSI treatment

Exclusion Criteria:

* Repeated implantation failures (with previous 3 or more IVF/ICSI failures)
* moderate to severe endometriosis
* untreated hydrosalpinx
* untreated endometrial disease
* contraindications for assisted reproductive techniques or gestation
* a history of ovarian surgery
* expected poor ovarian response (POR) or previous POR
* polycystic ovarian syndrome
* participants in clinical trials of other drugs within one month prior to enrollment; • hypersensitivity to follicle-stimulating hormone α, FSH, human menopausal gonadotropin, LH or excipients
* uncontrolled endocrine diseases (such as hyperthyroidism, hypothyroidism, adrenal gland disease, obesity, etc.)
* percutaneous epididymal sperm aspiration or testicular sperm aspiration

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate at 12 weeks' gestation | At 12 weeks' gestation
  Gestational sac with embryocardia-beat detected on ultrasound at 12 weeks' gestation

SECONDARY OUTCOMES:
Number of retrieved oocytes | Two weeks after oocyte retrieval
  Total number of retrieved oocytes

OTHER OUTCOMES:
The normal fertilization rate | Two weeks after oocyte retrieval
  The rate of fertilization with two pronuclear
The rate of high quality embryos | Two weeks after oocyte retrieval
  Number of high quality embryos / number of normal fertilized and cleavaged embryos
Implantation rate | Four to five weeks after embryo transfer
  Number of gestational sac / number of transferred embryos
Clinical pregnancy rate | Four to five weeks after embryo transfer
  Gestational sacs detected on ultrasound four to five weeks after embryo transfer
early miscarriage rate | At 12 weeks' gestation
  Misscarriage within 12 weeks' gestation

CONTACTS AND LOCATIONS:
Overall Officials: Dongzi Yang, doctor, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Hui Chen, doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Ruiqi Li, doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Xiaoli Chen, doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Lin Li, doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Ping Pan, doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Jia Huang, doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT05412147/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT05412147/ICF_001.pdf